CLINICAL TRIAL: NCT02789358
Title: A Time-to-effect Based Dosing Strategy in Cryoballoon Ablation of Patients With Paroxysmal Atrial Fibrillation. Results of the the plusONE Randomized Multicenter Trial
Brief Title: A Time-to-effect Based Dosing Strategy in Cryoballoon Ablation of Patients With Paroxysmal Atrial Fibrillation
Acronym: plusONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Principal Investigator, Angel Ferrero, MD-PhD, Fundación para la Investigación del Hospital Clínico de Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FIHCValencia
Record Dates: First submitted 2016-05-17; First posted 2016-06-03 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Atrial Fibrillation
Keywords: cryotherapy
MeSH Terms: conditions — Atrial Fibrillation | interventions — Adenosine Triphosphate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Arm (Active Comparator): Conventional protocol for cryoablation:
  At least 2 applications of 180s each
  Interventions: Other: Conventional cryotherapy dosage; Device: Arctic Front Advance ST Cryoenergy Balloon Catheter; Drug: Adenosine triphosphate; Device: nECG platform Nuubo®
- Study Arm (Experimental): Experimental protocol for cryoablation:
  Time to effect + 1 minute and a bonus application of 120s
  Interventions: Other: Experimental cryotherapy dosage; Device: Arctic Front Advance ST Cryoenergy Balloon Catheter; Drug: Adenosine triphosphate; Device: nECG platform Nuubo®

INTERVENTIONS:
Other: Conventional cryotherapy dosage — Cryotherapy dosage: 180 seconds applications until block of the pulmonary vein plus 1 bonus freezing of 180 seconds
  Arms: Control Arm
Other: Experimental cryotherapy dosage — cryotherapy dosage: applications "time to block of the vein" plus 60 seconds long until block of the vein plus 1 bonus freezing of 120 seconds
  Arms: Study Arm
Device: Arctic Front Advance ST Cryoenergy Balloon Catheter — Electrical isolation of pulmonary veins with Arctic Front Advance cryoballoon
Drug: Adenosine triphosphate — 12 mg of adenosine triphosphate are administrated intravenously to test dormant conduction in pulmonary veins apparently disconnected
Device: nECG platform Nuubo® — 30 days electrocardiographic monitoring system to detect atrial fibrillation episodes after ablation

SUMMARY:
This study aims to validate a new dosage of cryotherapy based on time to effect in pulmonary vein ablation procedures in patients with paroxysmal atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least 2 documented episodes of paroxysmal Atrial Fibrillation (AF) which are not responders to at least one antiarrythmic drug

Exclusion Criteria:

* Previous left atrial ablation procedure or surgery
* left atrium diameter > 50mm
* presence of intracardiac thrombus
* Left ventricular ejection fraction < 40%
* Heart failure class III-IV
* Severe valvulopathies
* Acute coronary syndrome or cardiac surgery within the previous 3 months of enrollment
* Transient ischemic attack/stroke within the previous 6 months of enrollment
* life expectancy less than 1 year
* Any contraindication to the procedure according to the current clinical practice

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-12; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation-free survival, without antiarrhythmic drug therapy | 12 months

SECONDARY OUTCOMES:
Mean number of cryotherapy applications per patient to complete isolation | Intraprocedural
Total cryotherapy time | Intraprocedure
  Total cryotherapy time of applications needed per patient
Time required to complete isolation of all the pulmonary veins (LA time) | Intraprocedure
  Time from the end of transeptal approach until the withdrawal of the cryoballoon
Total procedure time | Intraprocedure
  Time from the local anesthesia is administrated until the whole procedure is finished
Acute reconnection of pulmonary veins | Intraprocedure
  Number of veins reconnected after a 30 minutes waiting period since the end of procedure and with adenosine test
Adverse events | Intraprocedure
  Number of participants with procedural-related adverse events as assessed by by CTCAE v4.0
Total number of atrial fibrillation episodes monitored by Nuubo system | 12 Months
Total time in atrial fibrillation monitored by Nuubo system | 12 months
  Total time in atrial fibrillation monitored by Nuubo system in hours
Atrial fibrillation burden detected by Nuubo system | 12 Months
  total time in atrial fibrillation related to the hole time of monitoring (percentage)

CONTACTS AND LOCATIONS:
Overall Officials: Ángel Ferrero De Loma-Osorio, MD, PhD, Principal Investigator — Cardiologist
Locations (1):
- Hospital Clínico Universitario de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferrero-de-Loma-Osorio A, Garcia-Fernandez A, Castillo-Castillo J, Izquierdo-de-Francisco M, Ibanez-Criado A, Moreno-Arribas J, Martinez A, Bertomeu-Gonzalez V, Lopez-Mases P, Ajo-Ferrer M, Nunez C, Bondanza-Saavedra L, Sanchez-Gomez JM, Martinez-Martinez JG, Chorro-Gasco FJ, Ruiz-Granell R. Time-to-Effect-Based Dosing Strategy for Cryoballoon Ablation in Patients With Paroxysmal Atrial Fibrillation: Results of the plusONE Multicenter Randomized Controlled Noninferiority Trial. Circ Arrhythm Electrophysiol. 2017 Dec;10(12):e005318. doi: 10.1161/CIRCEP.117.005318. PMID 29247029